CLINICAL TRIAL: NCT04426162
Title: Effects of Memory Boot Camp on Brain Function in Adults With Symptoms of Mild Cognitive Impairment (MCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurocore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-127
Record Dates: First submitted 2020-05-13; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Memory Boot Camp Participants (Experimental): All subjects undergo a 12-week control period, followed by a multi-domain 12-week memory program.
  Interventions: Other: Multi-domain Intervention

INTERVENTIONS:
Other: Multi-domain Intervention — Intervention includes neurofeedback, heart rate variability biofeedback, memory and cognitive training, and one-on-one coaching to encourage behavior change in diet, sleep, physical fitness, and stress reduction.

SUMMARY:
This is a prospective controlled clinical trial to determine the effects of a 12-week Memory Boot Camp (MBC) program on cognitive function in older adults with symptoms of Mild Cognitive Impairment.

DETAILED DESCRIPTION:
This prospective trial evaluates the 12-week, multi-domain Memory Boot Camp program for adults ages 55 to 85 with symptoms of mild cognitive impairment. The Memory Boot Camp program incorporates neurofeedback, heart rate variability biofeedback, memory and cognitive training, and one-on-one coaching to encourage behavior change in diet, sleep, physical fitness, and stress reduction. Participants are evaluated via neurocognitive assessments, questionnaires, quantitative electroencephalography parameters, and heart rate variability parameters at four time points: baseline, pre-program, post-program, and follow-up. The trial included a 12-week waiting period between baseline and pre-program, such that each participant acts as their own control, and follow-up takes place six months after completion of the program.

ELIGIBILITY:
Inclusion Criteria:

* Subjective memory concerns
* At least a high school education
* Having a current primary care doctor (or agreement to get a primary care doctor)
* Ability to read and write English
* Time availability of 4-5 hours/week
* Be in good general health

Exclusion Criteria:

* Major depression
* Known neurological illness (e.g. Alzheimer's or other dementia, Parkinson's, epilepsy, multiple sclerosis)
* Serious psychiatric diagnosis
* Substance abuse
* Complete blindness or deafness
* Plans to be out of town for more than 10 days during the active phase of the trial
* Current or past client of the Sponsor
* Complete blindness or deafness
* Employee or family member of Sponsor employee

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) | Baseline (Month 0), program start (Month 3), program completion (Month 6), and 6-month post-program follow-up (Month 12).
  The MoCA is a validated, brief assessment tool that measures MCI and is widely used. Individuals are scored on seven different domains: visuospatial/executive, naming, attention, language, abstraction, delayed recall, and orientation.

OTHER OUTCOMES:
Change in Neurotrax BrainCare Testing Suite | Baseline (Month 0), program start (Month 3), program completion (Month 6), and 6-month post-program follow-up (Month 12).
  Neurotrax was originally developed and validated for the diagnosis of MCI in clinical practice and in research (at that time it was called "Mindstreams"). Neurotrax has been further validated since then in both demented and normally-aging populations.There are 7 domains covered by this series of tests: Memory, Executive Function (Thinking), Attention, Visual Spatial, Verbal Function, Problem Solving and Working Memory.
Change in Beck Depression Inventory-II (BDI) | Baseline (Month 0), program start (Month 3), program completion (Month 6), and 6-month post-program follow-up (Month 12).
  The BDI is a twenty-one item self-report inventory, and one of the most widely used instruments for measuring severity of depression.
Change in Beck Anxiety Inventory (BAI) | Baseline (Month 0), program start (Month 3), program completion (Month 6), and 6-month post-program follow-up (Month 12).
  The BAI is a twenty-one item self-report inventory, and is a widely-used instrument for measuring subjective, somatic, or panic-related symptoms of anxiety.
Change in Insomnia Severity Index (ISI) | Baseline (Month 0), program start (Month 3), program completion (Month 6), and 6-month post-program follow-up (Month 12).
  The ISI is a 7-item self-report inventory. The questionnaire is designed to assess the subject's sleep patterns and presence of or severity of insomnia during a 14-day period.
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline (Month 0), program start (Month 3), program completion (Month 6), and 6-month post-program follow-up (Month 12).
  The PSQI is a 19-item self-report inventory. The survey is designed to measure sleep quality and disturbances over a one-month interval in clinical populations. The nineteen items generate a global score as well as seven component scores (subjective sleep quality; sleep latency; sleep duration; habitual sleep efficacy; sleep disturbances; use of sleeping medication; daytime dysfunction).
Change in Work and Social Adjustment Scale (WSAS) | Baseline (Month 0), program start (Month 3), program completion (Month 6), and 6-month post-program follow-up (Month 12).
  The WSAS is a five-item self-report inventory, which provides a measure of global functional impairment, due to memory concerns.
Change in Quantitative Electroencephalography (QEEG) | Baseline (Month 0), program start (Month 3), program completion (Month 6), and 6-month post-program follow-up (Month 12).
  EEG activity will be collected 19 electrode locations, according to standard 10-20 site placement standards. Information about EEG absolute and relative power from 1 - 30 Hz will be collected at every location, as well as pairwise combinations of coherence and phase measures.Data will be compared to the Neuroguide age-normed QEEG database.
Change in Heart Rate Variability (HRV) | Baseline (Month 0), program start (Month 3), program completion (Month 6), and 6-month post-program follow-up (Month 12).
  HRV parameters include mean heart rate and two common time-domain measures used to calculate HRV: the standard deviation of normal to normal beat intervals (SDNN) and the root mean square of successive normal to normal beat interval differences (RMSSD).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Neurocore Brain Performance Center, Boca Raton, Florida
  - Neurocore Brain Performance Center, Palm Beach Gardens, Florida
  - Neurocore Brain Performance Center, Grandville, Michigan